CLINICAL TRIAL: NCT00484744
Title: Acetaminophen Versus Ibuprofen for the Control of Immediate and Delayed Pain Following Orthodontic Separator Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 07 04-054
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Orthodontic Pain
Keywords: pain; orthodontic; acetaminophen; ibuprofen; separator
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Cellulose; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acetaminophen (Experimental)
  Interventions: Drug: Acetaminophen
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen
- Avicel (Placebo Comparator)
  Interventions: Drug: Avicel (placebo)

INTERVENTIONS:
Drug: Acetaminophen
  Arms: Acetaminophen
Drug: Avicel (placebo)
  Arms: Avicel
Drug: Ibuprofen
  Arms: Ibuprofen

SUMMARY:
The purpose of this research study is to compare pain control effectiveness of two medicines and a placebo (a dummy pill that does not contain any pain relieving medication) to see which one works better at preventing pain when taken both 1 hour before and 6 hours after orthodontic separators are placed. The research hypothesis is that there will be a significant difference in pain as measured by Visual Analogue Scales (VAS) over time and that this effect will differ for acetaminophen versus ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic treatment requires banding of posterior teeth
* Orthodontic treatment requires the placement of two or more separators
* Able to swallow analgesic pills
* English speaking
* Age 9-17
* Minimum weight requirement of 88 pounds

Exclusion Criteria:

* Orthodontic appliances are present in the mouth
* Use of acetaminophen or ibuprofen is contraindicated (allergy, GI problems)
* Antibiotics or analgesics are currently in use
* History of systemic disease exists (arthritis, diabetes, cystic fibrosis)
* Significant cognitive impairment

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pain/discomfort levels reported on Visual Analogue Scales | Assessments conducted at six intervals during a 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Shelliann A Kawamoto, DDS, Principal Investigator — University of Missouri-Kansas City School of Dentistry Department of Orthodontics and Dentofacial Orthopedics; Karen Williams, RDH, MS, PhD, Study Chair — University of Missouri-Kansas City School of Dentistry
Locations (2):
- United States (2):
  - Orthodontic office of Drs. Dan Blackwell, Beth Blackwell-Nill, Scott Francois, Lee's Summit, Missouri
  - Orthodontic office of Dr. James Osborne, Lee's Summit, Missouri